CLINICAL TRIAL: NCT04176432
Title: Mortality and Complications After Emergency Laparotomy in Patients 80 Years Old or Older
Brief Title: Survival After Emergency Laparotomy in Octogenarians
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/610; REK 9526 (Other: Regional Ethics Committe)
Record Dates: First submitted 2019-09-27; First posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Abdomen, Acute; Surgery--Complications; Postoperative Complications; Frailty
Keywords: Emergency surgery; Frailty; Elderly; Postoperative complications
MeSH Terms: conditions — Abdomen, Acute; Postoperative Complications; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Other: No intervention — Retrospective observational study with no intervention

SUMMARY:
In this single-center retrospective study we wanted to investigate mortality and postoperative complications after emergency laparotomy performed in patients aged 80 years or above.

DETAILED DESCRIPTION:
Methods:

During 2015-2016 106 patients aged 80 years or above underwent emergency laparotomy at Haukeland University Hospital.

Primary outcome was mortality at 30 days. Secondary outcomes were mortality at 90 days, 1 year, postoperative complications and level of care at discharge.

The Medical records were reviewed in detail and mortality and postoperative morbidity were registered. Post-operative complications were defined according to the European Perioperative Clinical Outcome (EPCO) definitions and included if they were Clavien Dindo grade 2 or above.

ELIGIBILITY:
Inclusion Criteria:

* emergency laparotomy in patients 80 years or above

Exclusion Criteria:

* palliative surgery
* abdominal surgery other than gastrointestinal
* abdominal surgery without midline incision

Min Age: 80 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients admitted to Haukeland University Hospital during 2015-2016
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Number of Deaths within 30 days after emergency laparotomy | From date of emergency laparotomy until 30 days after surgery
  Mortality at 30 days after date of emergency laparotomy

SECONDARY OUTCOMES:
Number of Deaths within 90 days after emergency laparotomy | 90 days after emergency laparotomy
  Mortality at 90 days after date of emergency laparotomy
Number of Deaths within 1 year after emergency laparotomy | 1 year after emergency laparotomy
  Mortality at 1 year after date of emergency laparotomy
Postoperative complications | Postoperative complications registered in medical records from date of emergency laparotomy until death in hospital or discharge from hospital, whichever came first.
  Number of patients having a postoperative complication as defined by the European Perioperative Clinical Outcome Definitions (EPCO) will be reported. The EPCO definitions state universal description of various common postoperative complications, like f.ex pulmonary complications, major adverse cardiac events, urinary tract infections and so on. This is a way of securing a universal approach to postoperative complications.
  We will grade complications according to the Clavien Dindo classification. According to this classification postoperative complications are graded from 1 to 5, where 1 indicates least severity of complication and 5 indicating worst severity. We will report number of patients having complications from grade 2 to grade 5.
Level of care at discharge | Up to 90 days from date of emergency laparotomy.
  From the medical records will be retreived information regarding dependency in activities of daily living (ADL) at discharge. Specifically will be measured number of patients discharged to own home, and number of patients discharged to nursing home facility. Also will be measured number of patients transferred to other hospital.